CLINICAL TRIAL: NCT00211419
Title: Pilot Study of the Combination of Anecortave Acetate 15mg Delivered by Posterior Juxtascleral Injection and Triamcinolone Acetonide 4mg Delivered by Intravitreal Injection for the Treatment of Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Study of the Combination of Anecortave Acetate and Triamcinolone Acetonide for the Treatment of Exudative Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Manhattan Eye, Ear & Throat Hospital (Other)
Collaborators: Alcon Research (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: Double Injection
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2005-09

CONDITIONS: Maculopathy, Age-Related
Keywords: Exudative Age-Related Macular Degeneration; AMD
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate; Triamcinolone; Photochemotherapy; Verteporfin

INTERVENTIONS:
Drug: Anecortave Acetate 15 mg
Drug: Triamcinolone Acetate 4 mg
Procedure: Photodynamic Therapy with Verteporfin
Procedure: Thermal Laser

SUMMARY:
The purpose of this study is to evaluate the safety of combining juxtasclerally administered anecortave acetate 15 mg with triamcinolone acetate 4 mg administered intravitreally following photodynamic therapy with verteporfin for the treatment of exudative age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

1. A male or female with evidence of exudative age-related macular degeneration with clinical/angiographic/optical coherence tomography (OCT) findings of subfoveal choroidal neovascularization (CNV) which has not responded to current therapy
2. Baseline best-corrected visual acuity (BCVA) 20/40 to 20/640
3. Patient must be willing and able to comply with the protocol and provide informed consent.

Exclusion Criteria:

1. Patients on intravenous, subcutaneous, or anticoagulant therapy (with the exception of aspirin and antiplatelet therapy) and cannot take a 5 day holiday from therapy prior to the injection procedure. Note: Patients on oral anticoagulant therapy may be considered to participate if the physician responsible for monitoring the anticoagulant therapy agrees that the patient may take a 5 day holiday from therapy prior to each anecortave injection. The attending doctor must notify the principal investigator and this notification will be made part of the source documentation. Anticoagulant therapy may resume either the evening of or the morning after the injection procedure.
2. Patient with known glaucoma or steroid induced ocular hypertension
3. Intraocular pressures of 21 mmHg or greater at time of entry into the study
4. Patient with significantly compromised visual acuity in the study eye due to concomitant ocular conditions
5. Patients who have undergone intraocular surgery within last 2 months or capsulotomy within last month in study eye
6. Patient participating in any other investigational drug study
7. Inability to obtain photographs to document CNV (including difficulty with venous access)
8. Concomitant oral steroids or topical ophthalmic steroid use
9. Sub-Tenon's injection of steroids within the past 6 months
10. Patient with significant liver disease or uremia
11. Patient with known adverse reaction to indocyanine green, iodine, verteporfin, or triamcinolone
12. Patient is pregnant or nursing
13. Age less than 50 years old

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Slakter, MD, Principal Investigator — Manhattan Eye, Ear & Throat Hospital
Locations (1):
- Manhattan Eye, Ear & Throat Hospital, New York, New York, United States